CLINICAL TRIAL: NCT05583175
Title: Study of Venetoclax and Reduced-intensity Conditioning Regimen(RIC) for Allogeneic Stem Cell Transplantation(Allo-HSCT) in Elderly Patients With High-risk Myeloid Malignancies
Brief Title: Venetoclax Plus RIC Regimen Allo-HSCT for Elderly Patients With High-risk Myeloid Malignancies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xianmin Song, MD (Other)
Responsible Party: Sponsor-Investigator, Xianmin Song, MD, Head of Hematology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-202202-VEN-RIC
Record Dates: First submitted 2022-10-09; First posted 2022-10-17 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Leukemia, Myeloid, Acute; MDS; Hematopoietic Stem Cell Transplantation; Myeloid Malignancy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax plus RIC (Experimental): Administration with oral Venetoclax plus RIC regimen for allo-HSCT in the elderly patients with myeloid malignancies.
  Interventions: Drug: Venetoclax plus RIC

INTERVENTIONS:
Drug: Venetoclax plus RIC — Eligible patients will receive Venetoclax plus RIC regimen allogeneic transplantation. The treatment regimen is: Venetoclax 100mg/d - 10d, 200mg/d - 9d (first use and NR or untreated MDS), 400mg/d, - 8d~ - 2d (7d); Fludarabine: 30mg/m2/d, - 6d~-2d (5d), Cytarabine: 1g/m2/d, - 6d~-2d (5d) Busulfan: 3.2mg/m2/d, - 6d~-5d (2d), TBI: 3 Gray, - 1d.

SUMMARY:
This study is a single center, single arm, prospective, phase II clinical study to evaluate the efficacy and safety of Venatoclax combined with reduced intensity conditioning regimen allo-HSCT in the treatment of high-risk myeloid malignancies in the elderly patients.

DETAILED DESCRIPTION:
Eligible patients will receive Venetoclax plus RIC regimen allogeneic transplantation. The treatment regimen is: Venetoclax 100mg/d - 10d, 200mg/d - 9d (first use and NR or untreated MDS), 400mg/d, - 8d~ - 2d (7d); Fludarabine: 30mg/m2/d, - 6d~-2d (5d), Cytarabine: 1g/m2/d, - 6d~-2d (5d) Busulfan: 3.2mg/m2/d, - 6d~-5d (2d), total body irradiation(TBI): 3 Gray, - 1d.

Primary end point: 1 year and 2 year progression free survival (PFS) after transplantation. Secondary end point: incidence of acute GVHD within 180 days after transplantation; cumulative rate of relapse, overall survival(OS), graft-versus-host disease (GVHD)-free relapse-free survival(GRFS), non-relapse mortality(NRM), and incidence of chronic GVHD at 1 and 2 years after transplantation; The reactivation rate of cytomegalovirus(CMV) and Epstein-Barr virus (EBV) within 1 year after transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 55 years old;
2. High risk myeloid malignancies： 1）No hematological remission(NR) after induction/re-induction treatment for AML; 2）Morphological remission but with persistent positive minimal resident disease(MRD) (Flow cytometry>0.01% and/or fusion gene positive and/or digital polymerase chain reaction(PCR) positive）; 3）High risk acute myeloid leukemia(AML) according to 2022 European Leukemia Net(ELN) risk stratification； 4）High risk myelodysplastic syndrome(MDS): IPSS-R score ≥ middle risk-2; therapy-related MDS; MDS with mutation of ASXL1, EZH2, RUNX1, SRSF2, U2AF1, STAG2, NRAS, ZRSR2, or TP53； 5）High risk chronic myelomonocytic leukemia(CMML), MDS/MPN.
3. Patients must have appropriate donor:

1）Related donor must be HLA-A, - B, - C, - DQB1 and - DRB1 matched at least 5/10; 2）Unrelated donor must be HLA-A, - B, - C, - DQB1 and - DRB1 matched at least 8/10; 4. Hematopoietic cell transplantation-comorbidity Index(HCT-CI) score ≤ 4。 5. Eastern Cooperative Oncology Group(ECOG) score 0-2。 6. Liver, kidney and cardiopulmonary functions meet the following requirements:

1. Creatinine≤1.5×ULN;
2. Left ventricular ejection fraction >50%;
3. Baseline oxygen saturation>92%;
4. Total bilirubin≤1.5×ULN；ALT and AST≤2.0×ULN；
5. DLCO≥ 40% and FEV1 ≥ 50%。 7. Able to understand and sign the Informed Consent Document.

Exclusion Criteria:

1. Patients with Venetoclax ineffectiveness;
2. Malignant tumors other than acute myeloid leukemia within 5 years prior to screening, in addition to adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, and ductal carcinoma in situ after radical resection；
3. ECOG socre>2;
4. HCT-CI score> 4。
5. Any instability of systemic disease, including but not limited to unstable angina, cerebrovascular accident, or transient cerebral ischemic (within 3 months prior to screening), myocardial infarction (within 3 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ III), need drug therapy of severe arrhythmia, liver, kidney, or metabolic disease; patients with pulmonary hypertension
6. Uncontrolled infection during screening period; Hemodynamic instability associated with infection,a new infection or aggravation of the original infection;new lesions on imaging;fever of unknown cause;
7. Patients with symptoms of central nervous system;greater than grade 2 requiring treatment,paralysis,aphasia,acute cerebral infarction,severe traumatic brain injury,schizophrenia;
8. HIV infection;
9. Patients with active hepatitis B virus (HBV) and active hepatitis C virus (HCV) need antiviral treatment; Patients at risk of HBV activation refer to patients with positive HBsAg or HBeAb but not receiving anti-HBV treatment;
10. History of autoimmune disease；
11. Pregnant or lactating women；
12. Fertile men and women who are unwilling to use contraceptive technology during the treatment period and within 12 months after treatment.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 1- year PFS
  Progression free survival for all patients enrolled
PFS | 2- year PFS
  Progression free survival for all patients enrolled

SECONDARY OUTCOMES:
OS | 1- year OS
  Overall survival for all patients enrolled
OS | 2- year OS
  Overall survival for all patients enrolled
aGVHD rate | 180 days after transplantation
  The incidence rate of acute GVHD after transplantation
cGVHD rate | 1 year after transplantation
  The incidence rate of chronic GVHD after transplantation
cGVHD rate | 2 years after transplantation
  The incidence rate of chronic GVHD after transplantation
Relapse rate | 1 year after transplantation
  Cumulative relapse rate after transplantation
NRM | 2 years after transplantation
  Non relapse mortality after transplantation
GVHD-free relapse-free survival(GRFS) | 2 years after transplantation
  Time from transplantation to the diagnosis of chronic GVHD or relapse
Reactivation rate of EBV and CMV | 1 year after transplantation
  Reactivation rate of Epstein-Barr virus and cytomegalovirus after transplantation
Reactivation rate of EBV and CMV | 2 years after transplantation
  Reactivation rate of Epstein-Barr virus and cytomegalovirus after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin Song, Principal Investigator — Shanghai General HospitalShanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia JS, Kim HT, Murdock HM, Cutler CS, Brock J, Gooptu M, Ho VT, Koreth J, Nikiforow S, Romee R, Shapiro R, Loschi F, Ryan J, Fell G, Karp HQ, Lucas F, Kim AS, Potter D, Mashaka T, Stone RM, DeAngelo DJ, Letai A, Lindsley RC, Soiffer RJ, Antin JH. Adding venetoclax to fludarabine/busulfan RIC transplant for high-risk MDS and AML is feasible, safe, and active. Blood Adv. 2021 Dec 28;5(24):5536-5545. doi: 10.1182/bloodadvances.2021005566. PMID 34614506